CLINICAL TRIAL: NCT01929759
Title: Advanced Neuroimaging Evaluation of the Central Nervous System Biological Changes Associated With Efavirenz Therapy and Switch to an Elvitegravir-based Regimen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Brigham and Women's Hospital (Other); Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Nina Lin, MD, Instructor in Medicine, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NeuroHIV001
Record Dates: First submitted 2013-08-23; First posted 2013-08-28 (Estimated); Results first posted 2017-07-28 (Actual); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: HIV Disease
Keywords: HIV; neurocognitive symptoms; efavirenz; elvitegravir; neurometabolites
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Elvitegravir, Cobicistat, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; elvitegravir; Cobicistat; Emtricitabine; Tenofovir

STUDY DESIGN:
Intervention Model Description: Treatment switch study
Oversight: Data Monitoring Committee: No

ARMS (1):
- Drug switching (Other): Single-arm with switch from baseline antiretroviral therapy with Atripla to Stribild for total of 8 weeks.
  Interventions: Drug: Stribild (elvitegravir, cobicistat, emtricitabine and tenofovir)

INTERVENTIONS:
Drug: Stribild (elvitegravir, cobicistat, emtricitabine and tenofovir) — Switch from Atripla (efavirenz, emtricitabine and tenofovir) to Stribild (elvitegravir, cobicistat, emtricitabine and tenofovir)for total of 8 weeks

SUMMARY:
In this study we will use a multi-modal imaging approach of MRS and fMRI to comprehensively assess the biological changes in the brain associated with EFV-based regimen (EFV/FTC/TDF), specifically alterations in the brain circuitry, function and local neurochemistry, and their correlation with neuropsychological function. In a cohort of HIV-infected patients who are clinically stable on the commonly use regimen of EFV/emtricitabine (FTC)/truvada (TDF) or Atripla, we propose to replace the EFV component with a new integrase inhibitor, elvitegravir (EVG) boosted with cobicistat (COBI), given as the EVG/COBI/FTC/TDF Single Tablet Regimen (STR) to evaluate the EFV-related neural alterations. This is a multidisciplinary study which involves a team of infectious disease experts in the field of HIV, neuroradiologists with expertise in fMRI and MRS techniques to study various central nervous system and psychiatric disorders and a psychiatrist with experience and expertise in research on abnormalities of affective and motivational processing in the context of neuropsychiatric disorders. We will utilize the established clinical research platform in the Infectious Disease outpatient clinical practice at the Brigham and Women's Hospital, where there is currently have many ongoing HIV-related studies and a large panel of HIV-infected patients motivated to be involved in clinically relevant research. We propose to use advanced neuroimaging to measure biologically changes in the brain associated with long-term EFV use with the following specific aims:

1. Determine changes in neurometabolites measured by MRS in the brain associated with long-term EFV use
2. Assess for alterations in neural activity correlated with affective symptoms associated with EFV vs STR use using fMRI, and their associations with changes in neurometabolites assessed by MRS, and with changes in cognition assessed by Trail Making and Digit Substitution Tests.
3. Determine changes in emotion, cognition and sleep quality after switching from EFV to STR, and how they correlate with subject treatment preference.

This clinical study will extend our current understanding of EFV neurotoxicity by further defining the nature of these biological changes. Further elucidation of the neurobiological underpinnings of EFV-induced CNS toxicity will have clinical relevance in improving the quality of life and drug adherence of HIV-infected patients on ART, especially among older patients or those with baseline neuropsychiatric disorders, whom at baseline are more vulnerable to neurocognitive decline from long-term HIV infection.

ELIGIBILITY:
Inclusion Criteria:

* Chronic HIV-infected individuals on suppressive regimen with EFV/FTC/TDF, for at least 6 months
* Undetectable HIV-1 RNA virus load for at least 6 months
* No co-infections with active hepatitis B and C
* Presence of at least moderate symptoms on 2 out of 3 subcores on the DASS
* No known active HIV-related and non-HIV related CNS infections
* Estimated glomerular filtration rate (EGFR) >60 ml/min
* Consent to switching to EVG/COBI/FTC/TDF
* Ages 18 - 65

Exclusion Criteria:

* History of CNS opportunistic infections or active CNS infections
* History of severe psychiatric disorder (excluding depression and anxiety)
* History of chronic neurological disorders, such as epilepsy or multiple sclerosis
* History of or current significant substance abuse or dependence and/or heavy alcohol use (>12 oz/wk)
* Any women who may be pregnant (positive urine pregnancy test or unprotected sex in 2 weeks prior to scan) or known to be pregnant
* Contraindications to undergoing fMRI, including metallic implants, claustrophobia, and medical conditions or medications that significantly affect cerebral blood flow or function.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Drug Switching
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Drug Switching
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 10
Baseline measures for Neurometabolites Based on MRS [Mean (Standard Deviation); unit: arbitrary units] — The arbitrary units are expressed as the output from MRS software. While similar to concentration (mM) due to assumptions in the software, it is best expressed as arbitrary units for comparison from baseline to the second time point.
  arbitrary units
    Posterior cingulate creatine | 19.09 (2.27)
    Posterior cingulate glutamate | 25.36 (3.73)
    Posterior cingulate GABA | 4.99 (1.29)
    Anterior cingulate creatine | 14.06 (2.44)
    Anterior cingulate glutamate | 19.16 (3.11)
    Anterior cingulate GABA | 4.21 (1.18)

OUTCOME MEASURES:

1. Primary Outcome: Change in Neurometabolites Based on Magnetic Resonance Spectroscopy (MRS)
Description: Assess the change in levels of neuro-metabolites measured by MRS from week 0 (before switching to the efavirenz-based therapy) and then at week 8 (after completing 9 weeks of integrase-inhibitor based regimen with Stribild). Two areas of the brain: 1) posterior cingulate gyrus and 2) anterior cingulate will be assessed for the levels of brain Cr, GABA and GLU.
Time Frame: week 0 to week 8
Population: The arbitrary units are expressed as the output from MRS software. While similar to concentration (mM) due to assumptions in the software, it is best expressed as arbitrary units for comparison from week 0 to week 8.
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | Drug Switching
Number analyzed (Participants) | 10
arbitrary units
  Posterior Cingulate Creatine | 19.61 (3.44)
  Posterior Cingulate Glutamate | 24.54 (3.69)
  Posterior Cingulate GABA | 6.71 (1.07)
  Anterior Cingulate Creatine | 12.08 (4.63)
  Anterior Cingulate Glutamate | 16.16 (6.00)
  Anterior Cingulate GABA | 3.67 (1.52)

2. Primary Outcome: Neural Activation Networks Using Functional Magnetic Resonance Imaging (fMRI)
Description: Assess changes in neural activation correlated with affective disturbances associated with efavirenz-based therapy using fMRI employing an Emotional Word/Go-NoGo task paradigm that probes affective symptomatologies typical with EFV use, specifically anxiety/dysphoria and affective dysregulation and their association with changes in cognitive function. Four brain regions of interests (ROIs) are specified to show the differential frontal-limbic activation patterns in the task-evoked neural responses to the 3 linear contrasts of Pre-switch / Post-switch / Pre- vs. Post-switch: [Negative Word vs. Neutral Word] x [No-Go Trial Block vs. Go Trial Block]: anterior Frontal Pole (aFP), posterior Cingulate Gyrus (pCG), dorsal anterior Cingulate Gyrus (daCG), Left Hippocampus (LHC). A linear mixed-effects model is utilized to examine the effect sizes of the key Regimen/Condition contrasts, with the Subject factor as the random-effect and Age incorporated as a co-variate of no interest.
Time Frame: week 0 and week 8
Population: 8 of 10 enrolled patients passed QA testing to be included in the final analyses. The 3 linear contrasts of Pre-switch/Post-switch/Pre- vs. Post-switch: [Neg vs.Neu] x [No-Go vs. Go] are reported as z-score (standardized effect size measures with SD=1). Z-score is obtained for each subject, group Z-score is obtained via a mixed-effects model.
Measure: Number; unit: z-score
Arm/Group | Drug Switching
Number analyzed (Participants) | 8
z-score
  PreVsPostXNegVsNeuXNoGoVsGo: aFP | 3.42
  PreVsPostXNegVsNeuXNoGoVsGo: pCG | 3.90
  PreVsPostXNegVsNeuXNoGoVsGo: daCG | -2.76
  PreVsPostXNegVsNeuXNoGoVsGo:LHC | -2.96
  Pre: NegVsNeuXNoGoVsGo: aFP | 3.39
  Pre: NegVsNeuXNoGoVsGo:pCG | 3.61
  Pre: NegVsNeuXNoGoVsGo: daCG | -3.15
  Pre: NegVsNeuXNoGoVsGo: LHC | -2.27
  Post: NegVsNeuXNoGoVsGo: aFP | -3.17
  Post: NegVsNeuXNoGoVsGo: pCG | -2.66
  Post: NegVsNeuXNoGoVsGo: daCG | 3.69
  Post: NegVsNeuXNoGoVsGo: LHC | 3.47

3. Secondary Outcome: Change in Other Neurometabolite Measured by MRS Between Week 0 and Week 8
Description: Use MRS to evaluate a fuller panel of known neurometabolites (in addition to the primary endpoints) between week 0 and week 8 to identify prominent and significant changes associated with EFV use.
Time Frame: week 0 to week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | Drug Switching
Number analyzed (Participants) | 10
arbitrary units
  Posterior cingulate glutathione | 5.06 (1.17)
  Posterior cingulate aspartate | 3.69 (0.98)
  Anterior cingulate glutathione | 3.17 (1.34)
  Anterior cingulate aspartate | 2.57 (1.29)

4. Secondary Outcome: Neurocognitive Changes
Description: Assess for changes in cognitive and affective function prior to and after switching off EFV-based regimen. Indexes used to access neurocognitive changes included:
  1. Wechsler Adult Intelligence Scale (WAIS-R) Digital Symbol Substitution Test: sensitive to brain damage, dementia, age and depressive changes. Range of 0-100, the higher the score the better the person's performance
  2. Hamilton Rating Scale for Depression (HAMD): Measure of depression. Score of 0-7 is normal, score of >20 is moderate/severe depression
  3. Depression Anxiety Stress Scale (DASS-21) the lower the score, the less severe depression, anxiety and stress. Scale range of 0-63
  4. Frontal Systems Behavior Scale (FRSBE): Increased score indicates greater behavioral impairment associated with frontal systems, range 37.2 to 186
  6. Spielberger state trait anxiety inventory (STAI): the higher the score the greater then anxiety level, range of 20 to 80.
Time Frame: week 0 and week 8
Population: Several Indexes were used to access neurocognitive changes: WAIS, HAMD, FRSBE, DASS-21, STAI.
  Participants were given these tests prior to and after drug switch.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Drug Switching
Number analyzed (Participants) | 10
units on a scale
  pre-switch WAIS | 49.3 (11.62)
  post-switch WAIS | 53.4 (12.60)
  pre-switch FRSBE | 77.5 (10.01)
  post-switch FRSBE | 70.4 (13.00)
  pre-switch HAMD | 5.5 (3.41)
  post-switch HAMD | 2.8 (2.20)
  pre-switch DASS depression | 7.6 (8.58)
  post-switch DASS depression | 3.4 (4.72)
  pre-swtich STAI | 28.8 (5.87)
  post-switch STAI | 24.2 (3.19)

5. Secondary Outcome: Fasting Lipid Profile
Description: Measure the change in fasting lipid panel prior to and after switching off EFV-based regimen.
Time Frame: 8 weeks
Population: Change in fasting lipid profile was measured: total cholesterol, HDL and LDL levels.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Drug Switching
Number analyzed (Participants) | 10
mg/dl
  pre-switch Total cholesterol | 178.8 (24.24)
  post-switch Total cholesterol | 168.5 (20.84)
  pre-switch HDL | 52.6 (16.49)
  post-switch HDL | 52.3 (19.42)
  pre-switch LDL | 106.1 (22.96)
  post-switch LDL | 97.4 (19.36)
  pre-switch triglyceride | 101.3 (50.39)
  post-switch triglyceride | 94.5 (30.50)

6. Secondary Outcome: Sleep Quality
Description: Assess for changes in sleep pattern and quality prior to and after switching off EFV-based regimen through a self-administered Pittsburg Sleep Quality Index (PSQI). Measure consists of 19 items with each weighted on 0-3 scale and the sum produces a total score, which ranges from 0-21. The lower the score the healthier the sleep quality; minimum Score = 0 (better); maximum Score = 21 (worse).
Time Frame: week 0 and week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Drug Switching
Number analyzed (Participants) | 10
units on a scale
  pre-switch PSQI index | 4.8 (2.30)
  post-switch PSQI index | 3.1 (1.66)

7. Secondary Outcome: ART Regimen Preference
Description: Evaluate patient preference in ART regimen (Atripla, EFV/FTC/TDF versus EVG/COBI/FTC/TDF) through a self-administered questionnaire.
Time Frame: week 0 and week 8
Population: Patients were surveyed at the end of the study with a single question regarding their ART preference. They are asked to pick one of the 3 answers: 1. prefer Atripla, 2. prefer the new drug (Stribild) or 3. no preference. The number of patients who would like to switch to study drug, Stribild, are indicated by the percentage.
Measure: Count of Participants; unit: Participants
Arm/Group | Drug Switching
Number analyzed (Participants) | 10
Participants
  Prefers Stribld | 9
  Prefers Atripla | 0
  No preference | 1

8. Secondary Outcome: Markers of Immune Activation
Description: Change in markers of immune activation and inflammation associated with change to Stibild: sCD14, IP-10,sCD163, IL-6)
Time Frame: week 0 and week 8
Population: Inflammatory markers were measured pre- and post-drug switch from Atripla to Stibild.
Measure: Mean (Standard Deviation); unit: pg/ML
Arm/Group | Drug Switching
Number analyzed (Participants) | 10
pg/ML
  pre-switch sCD14 | 3329000 (566684)
  post-switch sCD14 | 2879000 (867793)
  pre-switch IP-10 | 237.3 (204.8)
  post-switch IP-10 | 224.2 (201)
  pre-switch sCD163 | 732000 (559000)
  post-switch sCD163 | 599500 (319200)
  pre-switch MCP-1 | 102.2 (68)
  post-switch MCP-1 | 91.39 (43.02)
  pre-switch IL-6 | 1.255 (0.5921)
  post-switch IL-6 | 1.301 (0.7115)
  pre-switch TNFR1 | 833.2 (222.1)
  post-switch TNFR1 | 878.1 (198.8)

9. Secondary Outcome: Effect of EFV and Its Metabolites
Description: Level of EFV (efavirenz) in Atripla and its two known metabolites known to cause cerebral side effects, 7-hydroxy (OH) EFV and 8-OH EFV, were measured in the plasma prior to switch off Atripla and after 8 weeks of RAL-based regimen (no EFV).
Time Frame: week 0 and week 8
Measure: Number; unit: participants
Arm/Group | Drug Switching
Number analyzed (Participants) | 10
participants
  Number with detectable 7-OH and 8-OH (pre-switch) | 10
  Number with detectable 7-OH and 8-OH (post-switch) | 0

ADVERSE EVENTS:
Arm/Group | Drug Switching
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

LIMITATIONS AND CAVEATS:
One participant did not have repeat fMRI because the pre-switch fMRI was not done correctly. The patient did not fully understand the tasks to be performed, therefore no repeat follow up fMRI was done without the comparator study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No